CLINICAL TRIAL: NCT02928289
Title: Multi-Center Prospective Randomized Controlled Study of the Safety and Effectiveness of the Sight Sciences VISCO™360 System in Canaloplasty vs Selective Laser Trabeculoplasty in the Reduction of IOP in Primary Open Angle Glaucoma
Brief Title: Safety and Effectiveness of the Sight Sciences VISCO™360 Versus SLT in Primary Open Angle Glaucoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Sight Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIGHTVISCO-001
Record Dates: First submitted 2016-10-06; First posted 2016-10-10 (Estimated); Results first posted 2025-09-24 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Open-Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- VISCO360 ab interno canaloplasty surgery (Active Comparator): Subjects randomized to this arm will undergo a surgical procedure in which the VISCO360 Viscosurgical System will be used to microcatheterize and viscodilate Schlemm's canal (i.e., canaloplasty).
  Interventions: Device: VISCO360 ab interno canaloplasty surgery
- Selective Laser Trabeculoplasty (SLT) (Active Comparator): Subjects randomized to this arm will undergo the SLT procedure.
  Interventions: Device: Selective Laser Trabeculoplasty (SLT)

INTERVENTIONS:
Device: VISCO360 ab interno canaloplasty surgery — 360 degrees of viscodilation of Schlemm's canal
  Arms: VISCO360 ab interno canaloplasty surgery
Device: Selective Laser Trabeculoplasty (SLT) — 360 degrees of selective laser trabeculoplasty
  Arms: Selective Laser Trabeculoplasty (SLT)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Sight Sciences VISCO™360 Viscosurgical System in reducing intraocular pressure (IOP) in adult, pseudophakic subjects with open-angle glaucoma.

DETAILED DESCRIPTION:
This is a randomized study comparing viscodilation with the VISCO360 device to selective laser trabeculoplasty. Subjects with mild to moderate primary open-angle glaucoma undergo IOP-lowering medication washout at baseline and at Month 12. Subjects will be followed through Month 24.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary open-angle glaucoma (POAG) in the study eye.
* Pseudophakic with Posterior Chamber IOL (PCIOL)
* Able and willing to attend follow up visits for two years post-operative
* Able and willing to sign informed consent

Exclusion Criteria:

* Phakia or aphakia
* Previous glaucoma procedure with or without an implantable glaucoma device (including incisional surgery, ALT, iridectomy/iridotomy, etc.) [Subjects with one prior SLT application (>3 months prior to screening) or prior ECP (performed > 12 months prior to screening) can be enrolled].
* Use of more than 3 ocular hypotensive medications (combination medications count as 2 medications)
* Diagnosis of acute angle closure, traumatic, congenital, malignant, uveitic, pseudoexfoliative, pigmentary or neovascular glaucoma
* Abnormal angle anatomy as determined by gonioscopy (e.g. peripheral anterior synechiae, rubeosis or other angle abnormalities)
* Participation in any clinical trial ≤ 30 days prior to screening

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Ripley, Study Director — Sight Sciences, Inc.
Locations (6):
- United States (6):
  - Vold Vision, Fayetteville, Arkansas
  - Coastal Vision Medical Group, Orange, California
  - Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - El Paso Eye Surgeons, El Paso, Texas
  - Ophthalmology Associates, Fort Worth, Texas

REFERENCES:
- [Derived] Rolim-de-Moura CR, Paranhos A Jr, Loutfi M, Burton D, Wormald R, Evans JR. Laser trabeculoplasty for open-angle glaucoma and ocular hypertension. Cochrane Database Syst Rev. 2022 Aug 9;8(8):CD003919. doi: 10.1002/14651858.CD003919.pub3. PMID 35943114

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-nine potential subjects provided written informed consent, however only 17 met eligibility criteria and were then randomized and treated.
Pre-assignment Details: Subjects provided informed consent at the Screening visit and if the screening eligibility criteria were met, underwent a washout of their intraocular pressure (IOP) lowering medication (generally 4 weeks) before returning for the baseline visit where diurnal IOP was measured. Subjects meeting the diurnall IOP criteria at the baseline visit were than randomized and treated.
Period: Overall Study
Arm/Group | VISCO360 ab interno canaloplasty surgery | Selective Laser Trabeculoplasty (SLT)
Started | 7 | 10
Completed | 0 | 0
Not Completed | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VISCO360 ab Interno Canaloplasty Surgery | Selective Laser Trabeculoplasty (SLT) | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.1 (6.7) | 74.7 (11.5) | 75.4 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 4 | 8 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 8 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 10 | 17
Diurnal Intraocular Pressure [Mean (Standard Deviation); unit: mm Hg] — Mean of the IOP taken using Goldmann tonometry at 3 diurnal timepoints and measured in mm Hg
  mm Hg | 25.8 (4.3) | 25.1 (2.5) | 25.4 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Diurnal IOP at 12 Months (Measured in mm Hg)
Description: The mean of the difference between the baseline DIOP and the 12 month DIOP for each subject. Measurements at baseline and 12 months are following wash-out of glaucoma medication.
Time Frame: 12 months
Population: Only seven (7) subjects, 3 in the VISCO360 group, and 4 in the SLT group had completed the Month 12 endpoint visit at the time the study was terminated for poor enrollment. One of the 4 subjects in the SLT group underwent a secondary glaucoma procedure (gel stent) at Day 266 so the 12 month DIOP was imputed as the Baseline DIOP (per the protocol analysis plan).
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | VISCO360 ab interno canaloplasty surgery | Selective Laser Trabeculoplasty (SLT)
Number analyzed (Participants) | 3 | 4
mm Hg | -5.2 (7.6) | -3.6 (3.3)

2. Secondary Outcome: Proportion of Subjects Achieving a ≥ 20% Change in Mean Diurnal IOP at 12 Months
Description: Measurement is performed at 12 months following wash-out of glaucoma medication and is the number of subjects with 12 month DIOP that is at least 20% lower than the baseline DIOP divided by the number of subjects and multiplied by 100.
Time Frame: 12 months
Population: Only seven (7) subjects, 3 in the VISCO360 group, and 4 in the SLT group had completed the Month 12 endpoint visit at the time the study was terminated for poor enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | VISCO360 ab interno canaloplasty surgery | Selective Laser Trabeculoplasty (SLT)
Number analyzed (Participants) | 3 | 4
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | VISCO360 ab interno canaloplasty surgery | Selective Laser Trabeculoplasty (SLT)
All-Cause Mortality (participants affected / at risk) | 1/7 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/7 | 2/10
Other Adverse Events (participants affected / at risk) | 1/7 | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VISCO360 ab interno canaloplasty surgery (N=7) | Selective Laser Trabeculoplasty (SLT) (N=10)
Ocular adverse event (Eye disorders) | 0 (0) | 1 (1) — IOP increase requiring intervention with SLT
non-ocular (Cardiac disorders) | 1 (1) | 0 (0) — Second-Degree Atrioventricular Block
non-ocular (Cardiac disorders) | 0 (0) | 1 (1) — transient ischemic attach
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VISCO360 ab interno canaloplasty surgery (N=7) | Selective Laser Trabeculoplasty (SLT) (N=10)
Ocular adverse events (Eye disorders) | 1 (1) | 0 (0) — IOP increase >= 10 mmHg vs. baseline IOP occurring at any visit
ocular adverse event (Eye disorders) | 0 (0) | 1 (1) — Need for secondary surgical intervention
non-ocular adverse event (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Bronchitis
non ocular adverse event (General disorders) | 0 (0) | 1 (1) — Headaches
ocular adverse event (Eye disorders) | 0 (0) | 1 (1) — IOP increase requiring management with systemic medication or with surgical intervention
ocular adverse event (Eye disorders) | 0 (0) | 1 (1) — dryness
non ocular adverse event (General disorders) | 0 (0) | 1 (1) — Worsening vertigo

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After Sponsor's publication of trial results, the Institution and Principal Investigator may publish the results of the Study generated by the Institution, subject to the obligations of the CTA, and prior approval of Sponsor in writing. The Institution shall furnish Sponsor with a written copy of any proposed publication or disclosure at least 60 days prior to submission for publication or disclosure. Sponsor may request changes or other measures to ensure the information is fairly stated.

DOCUMENTS (2):
  • Study Protocol (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT02928289/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT02928289/SAP_001.pdf